CLINICAL TRIAL: NCT02920125
Title: A Study to Evaluate the Results of Integrative Treatment (by Including Ayurvedic Capsules Suved & Reimmugen) for Vascular Disease: Namely: Cerebro Vascular Accident - Embolic and Atherosclerotic, CVA, CAD, IHD,DVT,
Brief Title: Study the Result of Ayurvedic SUVED & Reimmugen (Colostrum) Treatment on Vascular Disease, CAD, CVA, DVT.
Acronym: SHARP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sujata Vaidya (Industry)
Collaborators: Smt. Kashibai Navale Medical College and General Hospital (Other); Health Solutions, India (Industry)
Responsible Party: Sponsor-Investigator, Sujata Vaidya, Researcher, Health Solutions, India
Organization: Health Solutions, India (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKNMC&GH-HS/001/2016; U1111-1187-7158 (Other: WHO)
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Cerebro Vascular Disease; Ischemic Heart Disease; Deep Vein Thrombosis; Peripheral Arterial Diseases; Vascular Disease
Keywords: Vascular disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Venous Thrombosis; Peripheral Arterial Disease; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Double Blind, Placebo controlled, two arm, on patients of vascular disease / atherosclerosis. Intervention is given in addition to ongoing conventional therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For subjects/patients -Control and Trial medication are packaged in same looking blister / alu alu strips.
  For Investigator and Outcome Assessor: no information on patient allocation (trial or Control group)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trial: Ayurvedic SUVED, REIMMUGEN (Active Comparator): Ayurvedic SUVED formulation comprises of 'Ghana' extract form; Dosage :3 months, 1 BD. Content: (500mg per capsule)Terminalia Arjuna: Withania somnifera; Terminalia chebula; Cyperus rotundus; Apium graveolens; Vitis vinifera; Piper longum; Fagonia Arabica; Emblica officinalis; Terminalia belerica; Nymphaea stellata; Punica granatum; Bacopa Monnieri; and stabilizing herbs.
  Reimmugen Cow-colostrum is a total natural product, used as nutritional supplement Dosage: 3months, 1 TDS Contents: IgA, IgE, IgM, IgG, IgD, PRPs, Lactoferrin, Transferrin, Interferons, Cytokines, Growth Factors (bFGF, vFGF, IGF I & II & Angiogenesis growth Factor, Endothelial growth Factor, Nerve growth factor, PDGF), natural Vitamins and Minerals.
  Interventions: Drug: SUVED; Combination Product: REIMMUGEN
- Control: grain flour (Placebo Comparator): Dummy medication in same packing to mask content given in same dose as active medication. Jowari and ragi flour used in capsules
  Interventions: Other: Grain flour placebo

INTERVENTIONS:
Drug: SUVED — Ayurvedic formulation in ghana (concentrated) in capsules; 500 mg each
  Other Names: Ayurvedic Suved
  Arms: Trial: Ayurvedic SUVED, REIMMUGEN
Combination Product: REIMMUGEN — Whole Cow colostrum in powder put in capsules; 300mg each
  Other Names: Reimmugen Cow Colostrum
  Arms: Trial: Ayurvedic SUVED, REIMMUGEN
Other: Grain flour placebo — Grain flour in capsules. Jowari flour in dummy Reimmugen and Ragi flour in dummy Suved placebos
  Arms: Control: grain flour

SUMMARY:
To evaluate the benefits of Ayurvedic SUVED & REIMMUGEN Colostrum for reduction/reversal of symptoms and study clinical progress in Vascular disease; CAD, CAV, Stroke, DVT patients.

DETAILED DESCRIPTION:
Aim: A non-invasive, effective, compatible, Integrative treatment option to address the growing burden of Vascular disease; Importance: Ayurvedic SUVED (cardio tonic, continuous clotlysis, endothelial repair, powerful rejuvenator, antioxidant) and Reimmugen (Cow Colostrum - IgG, GF) provides sustained Functional, symptomatic relief with clinical reports of regression of disease. No adverse interactions reported.

Application: Addition of SUVED & REIMMUGEN helps in:

* Acute MI, Thrombotic stroke, DVT, hastens symptomatic recovery, reduces hospitalization time, mortality, helps dissolve clots / soft thrombus; reversal of atherosclerotic plaques; improves functional life
* Improvements in Cardiac Function : LVEF; Global perfusion
* Rejuvenation of endothelium, vascular function.
* Improved physical strength: digestion; GI function; immunity; accelerated internal healing
* Secondary prevention to avoid incidences in post event treatment.

Health condition/problem studied Vascular disease, esp CVA, IHD, CAD, DVT, PAD Volunteers taken from OPD and IPD of SKNMC & GH with prior consent for participation.

Intervention is Medicament based given in addition to conventional ongoing therapy under the guidance of SKNMC doctors.

Study type Clinical trial: Double Blind placebo controlled trial. Interventional Trial: regular treatment. Evaluation of additional Integrative esp Ayurvedic medicaments on clinical and functional outcome.

Intervention and comparator agent

1. Ayurvedic ghana formulation named SUVED.
2. Whole Cow Colostrum called Reimmugen These will be given for a period of three months in addition to ongoing medication to study the additional benefit to patient in their functional and clinical investigations.

The control intervention/s is/are the interventions against which the study intervention is evaluated as double blind placebo.

Suved 1 BD for 3 months Reimmugen 1 TDS for 3 months In acute cases Suved 1 TDS Reimmugen 2 TDS for 3 months. Inclusion/ Exclusion criteria Inclusion criteria

Adult males or females with a diagnosis of Vascular disease leading to IHD, CAD, CVA, DVT, PAD at any stage.

Exclusion Criteria:

Pregnant and lactating women, Patients below age of 18 Acute IPD operative condition Patients undergoing interventional procedures / surgical treatments other than for Vascular disease; until they are discharged from intensive care; Haemorrhagic cerebro vascular stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females with a diagnosis of Vascular disease leading to IHD, CAD, CVA, DVT, PAD at any stage

Exclusion Criteria:

* Pregnant and lactating women
* Patients below age of 18
* Acute IPD operative condition
* Patients undergoing intervention procedures / surgical treatments other than for Vascular disease; until they are discharged from intensive care; Hemorrhagic cerebro vascular stroke

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
changes in IMT as a indicator of atherosclerosis reversal | 3 months active treatment
  Restoration of carotid IMT to non pathological state, supported with positive changes in functionality, relief from associated symptoms during treatment period of 3 months.

SECONDARY OUTCOMES:
Assessing the development/risk of ischaemic events in other circulations | 3 months
  Secondary outcomes assessing the development/risk of ischaemic events in other circulations. Eg; in a stroke patient, evaluation of coronaries.
  Evaluations done within the study period of 3 months for each patient.
  To study the occurance of new events in other territory.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shreepad M Bhat, MD, Principal Investigator — Smt Kashibai Navle Medical College & Gen Hospital
Locations (1):
- Smt Kashibai Navle Medical College and General Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
May share Data with other research agencies, Health Ministry or others.